CLINICAL TRIAL: NCT02696837
Title: Safety Control Study in Pediatric Inguinal Hernia Repair: Are Muscle Relaxants Necessary? Endotracheal Intubation vs Laryngeal Mask Airway
Brief Title: Pediatric Inguinal Hernia Repair: Are Muscle Relaxants Necessary? Endotracheal Intubation vs Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Collaborators: Pendik State Hospital (Unknown); Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., Principle Investigator, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PIRS002
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Inguinal Hernia; Endotracheal Intubation; Laryngeal Mask; Muscle Relaxants
MeSH Terms: conditions — Hernia, Inguinal; Muscle Hypotonia | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ETT & Muscle Relaxant (Active Comparator): Children undergoing laparoscopic inguinal hernia repair using PIRS method with Endotracheal Intubation and Muscle Relaxant
  Interventions: Device: ETT; Drug: Rocuronium
- ETT & No Muscle Relaxant (Active Comparator): Children undergoing laparoscopic inguinal hernia repair using PIRS method with Endotracheal Intubation and No Muscle Relaxant
  Interventions: Device: ETT; Other: No Muscle Relaxant
- Proseal LMA & No Muscle Relaxant (Active Comparator): Children undergoing laparoscopic inguinal hernia repair using PIRS method with Proseal Laryngeal Mask Airway and NO Muscle Relaxant
  Interventions: Device: Proseal LMA; Other: No Muscle Relaxant
- Proseal LMA & Subparalytic Muscle Relaxant (Active Comparator): Children undergoing laparoscopic inguinal hernia repair using PIRS method with Proseal Laryngeal Mask Airway and subparalytic dose Muscle Relaxant
  Interventions: Device: Proseal LMA; Drug: Rocuronium

INTERVENTIONS:
Device: ETT
  Arms: ETT & Muscle Relaxant; ETT & No Muscle Relaxant
Device: Proseal LMA
  Arms: Proseal LMA & No Muscle Relaxant; Proseal LMA & Subparalytic Muscle Relaxant
Drug: Rocuronium
  Arms: ETT & Muscle Relaxant
Other: No Muscle Relaxant
  Arms: ETT & No Muscle Relaxant; Proseal LMA & No Muscle Relaxant
Drug: Rocuronium
  Arms: Proseal LMA & Subparalytic Muscle Relaxant

SUMMARY:
In prospective, safety-control study; children undergoing laparoscopic inguinal hernia repair using PIRS (Percutaneous Internal Ring Suturing) method will be randomly assigned into four groups. Gr 1: Endotracheal intubation and muscle relaxant, Gr 2: Endotracheal Intubation without muscle relaxant, Gr 3: Proseal Laryngeal Mask Airway without muscle relaxant, Gr 4: Proseal Laryngeal Mask Airway with subparalytic does muscle relaxant. Apart from standard monitorization, all patients' intragastric pressures will also be monitored. Patients' age at presentation, gender, time of surgery, time of anesthesia, intragastric pressure, intraabdominal pressure, intraoperative findings and complications will be noted and compared between groups.

DETAILED DESCRIPTION:
In this prospective, safety-control study; children undergoing laparoscopic inguinal hernia repair using PIRS (Percutaneous Internal Ring Suturing) method will be randomly assigned into four groups.

Gr 1: Endotracheal intubation and muscle relaxant, Gr 2: Endotracheal Intubation without muscle relaxant, Gr 3: Proseal Laryngeal Mask Airway without muscle relaxant, Gr 4: Proseal Laryngeal Mask Airway with subparalytic does muscle relaxant.

Apart from standard monitorization, all patients' intragastric pressures will also be monitored. Patients' age at presentation, gender, time of surgery, time of anesthesia, intragastric pressure, intraabdominal pressure, intraoperative findings and complications will be noted and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years
* Diagnosed with inguinal hernia or communicating hydrocele
* Due to undergo laparoscopic inguinal hernia repair

Exclusion Criteria:

* Previous abdominal surgery
* Comorbidities that will effect surgical time, time under anesthesia, intragastric pressure and abdominal pressure

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Surgery Time | Intraoperative
  Time from skin prep to last suture
Time Under Anesthesia | Intraoperative
  Time from induction to moderate Alderete score of 9 or above
Intragastric Pressure | Intraoperative continuous monitoring
Intraabdominal Pressure | Intraoperative continuous monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, M.D., Principal Investigator — Maltepe University
Locations (1):
- Maltepe University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas DT, Gocmen KB, Tulgar S, Boga I. Percutaneous internal ring suturing is a safe and effective method for the minimal invasive treatment of pediatric inguinal hernia: Experience with 250 cases. J Pediatr Surg. 2016 Aug;51(8):1330-5. doi: 10.1016/j.jpedsurg.2015.11.024. Epub 2015 Dec 11. PMID 26777889
- [Result] Ozdamar D, Guvenc BH, Toker K, Solak M, Ekingen G. Comparison of the effect of LMA and ETT on ventilation and intragastric pressure in pediatric laparoscopic procedures. Minerva Anestesiol. 2010 Aug;76(8):592-9. Epub 2010 Jun 18. PMID 20661199
- [Result] Aydogmus MT, Turk HS, Oba S, Unsal O, Sinikoglu SN. Can Supreme laryngeal mask airway be an alternative to endotracheal intubation in laparoscopic surgery? Braz J Anesthesiol. 2014 Jan-Feb;64(1):66-70. doi: 10.1016/j.bjane.2012.12.008. Epub 2013 Dec 3. PMID 24565391
- [Result] Chen BZ, Tan L, Zhang L, Shang YC. Is muscle relaxant necessary in patients undergoing laparoscopic gynecological surgery with a ProSeal LMA? J Clin Anesth. 2013 Feb;25(1):32-5. doi: 10.1016/j.jclinane.2012.06.004. Epub 2012 Nov 2. PMID 23122973
- [Result] Liu HC, Tao WK, Zeng RF, ShangGuang WN, Li J, Huang WG, Dong ZL, Wang X, Lian QQ. Dose requirements of remifentanil for intubation in nonparalyzed Chinese children. Paediatr Anaesth. 2014 May;24(5):505-9. doi: 10.1111/pan.12354. Epub 2014 Feb 7. PMID 24708453